CLINICAL TRIAL: NCT00866710
Title: Behavioral Therapy to Treat Urinary Incontinence in Parkinson's Disease
Acronym: BETTUR PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlanta VA Medical Center (U.S. Federal Agency)
Collaborators: The John A. Hartford Foundation (Other)
Responsible Party: Principal Investigator, Camille Vaughan, MD, Investigator, Staff Physician, Atlanta VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6-38941
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Urinary Incontinence; Parkinson's Disease
MeSH Terms: conditions — Urinary Incontinence; Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Exercise-based behavioral therapy — Participants will be taught pelvic floor muscle exercises as well as urge suppression strategies to overcome the urge to void. In the first 20 participants, computer-assisted biofeedback will also be utilized to help participants identify the pelvic floor muscles and contract and relax these muscles while keeping the abdominal muscles relaxed

SUMMARY:
Background: Parkinson's disease affects up to 3% of persons over the age of 65. Lower urinary tract symptoms are a frequent cause of diminished quality of life in elderly persons and occur in up to 40% of persons with Parkinson's disease. While the exact mechanisms have not been determined, detrusor hyperactivity (hyperactivity of the bladder muscle) leading to symptoms of overactive bladder and urge incontinence is common. Behavioral and exercise-based therapies have relatively no side effects and have been shown to be an effective treatment for urge symptoms of overactive bladder in the aged population.

Hypothesis and Specific Aims: Behavioral therapy using pelvic floor muscle exercises will result in a 50% decrease in the number of incontinence episodes in elderly persons (age > 50) with Parkinson's disease. The specific aims for this pilot study include the following:

1. Complete a course of behavioral therapy using computer-assisted biofeedback in 20 subjects with UI associated with PD and determine how many potential subjects need to be screened and enrolled to achieve this sample size.
2. Determine the proportion of these patients who achieve a 50% or greater reduction in UI episodes.
3. Examine whether responsiveness is associated with characteristics of the Parkinson's disease, in particular disease severity as measured by the Unified Parkinson's Disease Rating Scale (UPDRS).
4. Assess the effectiveness of behavioral therapy without the use of computer-assisted biofeedback instruction in 10 additional subjects with PD and UI.

Methods: The first 20 participants will be enrolled in an 8-week treatment trial of behavioral therapies and pelvic floor muscle exercises with computer-assisted biofeedback. Ten additional participants will be enrolled in the 8-week treatment trial of behavioral therapy, but will not have computer-assisted biofeedback. Voiding diaries as well as urinary symptom and quality of life questionnaires will be used to assess response.

If persons with Parkinson's disease can complete the treatment trial and achieve a reduction in episodes of urinary incontinence with behavioral techniques this would lay the foundation for a larger, placebo-controlled trial. Assessment of responsiveness associated with severity of Parkinson's disease would also provide important information about the utility of this treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's disease
* ≥4 weekly episodes of UI with >50% of accidents associated with feelings of urgency where urgency is defined as the complaint of a sudden compelling desire to pass urine, which is difficult to defer
* Willingness to attend clinic visits
* Willingness to keep bladder diaries

Exclusion criteria:

* Cognitive impairment, as evidenced by a Folstein mini-mental status examination (MMSE) of < 24, or inability to produce an interpretable 7-day bladder diary
* Use of an indwelling urinary catheter
* Suggestion of bladder outlet obstruction as evidenced by having been prescribed in-and-out catheterization in the past 12 months, having a post-void residual by bladder ultrasound of ≥300 milliliters or a peak voiding flow rate of ≤ 4 mL/min on a void ≥ 125 mL in volume
* Severe uterine prolapse past the vaginal introitus
* Poorly controlled diabetes defined by a hemoglobin A1c (HgbA1c) of >8.0%
* Chronic renal failure and on hemodialysis
* Poorly controlled congestive heart failure or poorly controlled chronic obstructive pulmonary disease as evidenced on physical exam
* Genitourinary cancer with ongoing surgical or external beam radiation treatment
* Any unstable health condition expected to result in hospitalization or death within in the next 3 months as determined by principal investigator.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Bladder diary | 1 week

SECONDARY OUTCOMES:
Quality of Life Questionnaire | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C Vaughan, MD, Principal Investigator — Birmingham/Atlanta VA Geriatric Research Education and Clinical Center & Emory University
Locations (1):
- Atlanta VA Medical Center, Atlanta, Georgia, United States